CLINICAL TRIAL: NCT03976869
Title: An Open-Label, Multi-Centre, Phase I Study to Assess the Pharmacokinetics, Pharmacodynamics and Safety of 2-Week Treatment With Inhaled AZD7594 in Adolescents (12 to 17 Years) With Asthma
Brief Title: A Study to Assess the Pharmacokinetics (PK), Pharmacodynamics (PD) and Safety of 2-Week Treatment With Inhaled AZD7594 in Adolescents (12 to 17 Years) With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3741C00012
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: glucocorticoid receptor (GR) modulator (SGRM); non-steroidal; Asthma; Adolescents
MeSH Terms: conditions — Asthma | interventions — velsecorat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): The study will include adolescent patients of 12 to 17 years of age, with subgroups of 12-14 years age and 15-17 years age.
  Interventions: Drug: AZD7594

INTERVENTIONS:
Drug: AZD7594 — During treatment period, AZD7594 (360 µg per day) will be administered as oral inhalation via dry powder inhaler or DPI (SD3FL inhaler).

SUMMARY:
This is an open-label, multi-centre, Phase I study to assess the PK, PD and safety of 2 week treatment with inhaled AZD7594 in adolescent patients with asthma.

The study is planned to be conducted at 4-10 study sites in the United States. The study intends to include 24 patients (12 to 17-year-old patients). For each patient, the duration of participation in the study will be approximately 5 to 7 weeks (37 to 52 days).

DETAILED DESCRIPTION:
This is an open-label, multi-centre, Phase I study to assess the PK, PD and safety of 2 week treatment with inhaled AZD7594 in adolescent patients with asthma.

The study is planned to be conducted at 4-10 study sites in the United States. Eligible 12 to 17-year-old patients with asthma controlled on Global Initiative for Asthma (GINA) step 2 medication (ie, low dose inhaled corticosteroid [ICS] or leukotriene receptor antagonist [LTRA]), as evidenced by an asthma control questionnaire (ACQ-5) score ≤1.5, will be asked to stop their ongoing asthma maintenance treatment. After a washout period (14 to 21 days), all patients with confirmed reversibility will start study treatment, consisting of inhalations of AZD7594 (360 µg, delivered dose, via dry powder inhaler [DPI]) once daily for 15 to 16 days.

The study intends to include 24 patients in order to have 18 evaluable patients, enrolled in equal proportion in the age group of 12 to 14 years (inclusive), and the age group of 15 to 17 years (inclusive), with at least 7 patients in each subgroup.

For each patient, the duration of participation in the study will be approximately 5 to 7 weeks (37 to 52 days)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF) prior to any study-specific procedures from patient's parents/legal guardians is required and signed and dated informed assent from the patient.
2. Patient must be 12 to 17 years of age inclusive, at the time of signing the ICF/assent.
3. A minimum of 6-month documented history of asthma treated (daily or intermittently) for at least 3 months before screening (Visit 1) with either low dose inhaled corticosteroid (ICS) monotherapy or leukotriene receptor antagonist (LTRA) monotherapy.
4. Pre-bronchodilator FEV1 ≥70% of the predicted normal value at screening (Visit 1).
5. An ACQ-5 score <1.5 at screening (Visit 1).
6. Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to screening (Visit 1).
7. Body mass index (BMI) above the 5th percentile for the patient's age and gender and a minimum weight of 30 kg at screening (Visit 1).
8. Male or female
9. Negative pregnancy test (urine or serum) for post-menarcheal female patients at screening (Visit 1).
10. Post-menarcheal female patients must be willing to use a highly effective method of contraception which results in a low failure rate (ie, less than 1% per year). Sexual abstinence will be accepted as an effective method of contraception, provided a discussion occurred between the subject and investigator to confirm this lifestyle.

    After the washout period, patients are eligible to enter the treatment period only if all of the following inclusion criteria apply:
11. Negative pregnancy test (urine or serum) for post-menarcheal female patients at baseline (Visit 4).
12. FEV1 increase of at least 12% and 200 mL from baseline 15 to 30 minutes after 400 μg salbutamol (or albuterol equivalent of 360 µg) documented in the patient's medical history within 6 months of Visit 1, or confirmed at Visit 1 or Visit 2. In 12 to 14-year-old patients (who are likely to have a smaller forced vital capacity), positive reversibility testing could be based solely on the relative post bronchodilator response (at least 12%).

Exclusion Criteria:

Patients are eligible to enter the washout period if none of the following exclusion criteria apply:

Medical conditions

1. Any clinically significant disease or disorder (eg, cardiovascular, pulmonary other than asthma, gastrointestinal, liver, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment, severe obesity including weight-related health problems) which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the result of the study, or the patient's ability to participate in the study.
2. Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, at screening (Visit 1), which, in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study.
3. Prolonged QT interval corrected using Fridericia's formula (QTcF) ≥440 msec based on ECG at screening (Visit 1) or pre-dose at Visit 4, or family history of long QT syndrome.
4. Prolonged PR interval (>180 msec for ≤16-year-old patients and >200 msec for >16 year old patients) at screening (Visit 1) or pre-dose at Visit 4.
5. Heart rate <50 beats per minute (bpm) or >110 bpm.
6. History of or current alcohol or drug abuse (including marijuana), as judged by the Investigator.
7. Patients who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) at screening (Visit 1).
8. Hospitalisation due to asthma exacerbation or asthma exacerbation within 1 month prior to screening (Visit 1).
9. Lower respiratory tract infection within 1 month prior to screening (Visit 1).

   Prior/concomitant therapy
10. Patient who, in the opinion of the Investigator, is unable to abstain from protocol-defined prohibited medications during the study.

    Prior/concurrent clinical study experience
11. Participation in another clinical study with an investigational drug administered in the last 3 months before Visit 1, or participation in a method development study (no drug) 1 month prior to Visit 1.

    Note: Participation is identified as the completion of a treatment related visit.
12. A definite or suspected personal history of intolerance or hypersensitivity to drugs and/or their excipients, judged to be clinically relevant by the Investigator.

    Other exclusions
13. Inability to perform the required spirometry assessments, to use the AZD7594 inhaler or the short-acting beta agonist (SABA) inhaler, or to undergo blood sampling.
14. Parent/legal guardian involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
15. Judgement by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
16. Previous enrolment in the present study.
17. For post-menarcheal female patients only - currently pregnant, breastfeeding, or planning to become pregnant during the study.

After the washout period, patients are eligible to enter the treatment period if none of the following exclusion criteria apply:

1. An ACQ-5 score ≥3 at Visit 4.
2. SABA use of ≥12 puffs/day for ≥3 consecutive days during the washout period.
3. An asthma exacerbation that required treatment with ICSs or systemic steroids during the washout period.
4. A <70% compliance in completing asthma symptom score during the last 7 days of the washout period (ie, <5 out of 7 days with both morning and evening assessments completed).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration at steady state (Cmax,ss) at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma
Minimum observed plasma concentration at steady state (Cmin,ss) at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma.
Observed trough plasma concentration at end of dosing interval (τ) (Ctrough) at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma
Time of maximum observed plasma concentration at steady state (tmax,ss) at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma.
Area under the plasma concentration-time curve over a dosing interval (τ) at steady state (AUCτ) at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma.
Area under the plasma concentration curve from time zero to 12 hours post-dose (AUC0-12) under plasma concentration at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma.
Apparent total body clearance after extravascular administration at steady state (CLss/F) at Day 15 as part of PK evaluation | Pre-dose and 15, 30 minutes, 2, 4, 6, 8, 12 hours post-dose at Day 15
  To assess the PK profile of AZD7594 at steady state following daily inhalations for 2 weeks in adolescent patients with asthma.

SECONDARY OUTCOMES:
Relative change from baseline in plasma cortisol area under the effect curve from time zero to 12 hours post-dose (AUEC0-12) on Day 15 as part of PD evaluation | Pre-dose and 2, 4, 6, 8, 12 hours post-dose at Day 15
  To evaluate the PD of AZD7594 following daily inhalations for 2 weeks in adolescent patients with asthma.
Change from baseline in morning trough forced expiratory volume in 1 second (FEV1) on Day 15 as part of PD evaluation | At screening, Day 1 (pre-dose and 5, 15, 60 minutes post dose), Day 15 (pre-dose) and at end of study
  To evaluate the PD of AZD7594 following daily inhalations for 2 weeks in adolescent patients with asthma.
Change from baseline in asthma control questionnaire (ACQ-5) on Day 15 as part of PD evaluation | At screening, Day 1 (pre-dose) and Day 15 (pre-dose)
  To evaluate the PD of AZD7594 following daily inhalations for 2 weeks in adolescent patients with asthma. ACQ-5 is a 5 item questionnaire that scores symptoms on a 0-6 scale (where 0=none/no symptoms and 6=worst symptoms) . The form is completed by the patient during visits.

OTHER OUTCOMES:
Number of patients with adverse events and abnormal findings in vital signs, clinical laboratory parameters, physical examination, and electrocardigram (ECG) | From screening to follow-up (7-14 days)
  To evaluate the tolerability and safety of inhaled AZD7594

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Rolling Hills Estates, California
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Bethesda, Maryland
  - Research Site, Kansas City, Missouri
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home